CLINICAL TRIAL: NCT00947297
Title: A Phase 3, Open-Label Study of the Safety of HPN-100 for the Long-Term Treatment of Urea Cycle Disorders (Treat UCD)
Brief Title: Study of the Safety of HPN (Hyperion)-100 for the Long-Term Treatment of Urea Cycle Disorders (Treat UCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-007
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorder; UCD; hyperammonemia; Buphenyl; Sodium Phenylbutyrate
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPN-100 (Experimental): Patients who were treated with HPN-100
  Interventions: Drug: HPN-100

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a triglyceride that has a similar mechanism of action as NaPBA. It is a liquid with minimal taste and odor. Three teaspoons of HPN-100 (~17.4 mL) delivers equivalent of PBA that 40 tablets of NaPBA do.
  Other Names: GT4P, Glyceryl tri-(4-phenylbutyrate)

SUMMARY:
This was a long-term safety study HPN-100 in urea cycle disorder (UCD) subjects. Subjects were assessed regularly for safety and control of their venous ammonia. Hyperammonemic events were characterized with respect to contributing factors, such as intercurrent illness, diet, and noncompliance with medication.

DETAILED DESCRIPTION:
This was a one year long-term safety study of HPN-100 in UCD subjects. Subjects were assessed regularly for safety and control of their venous ammonia. Hyperammonemic events were characterized with respect to contributing factors, such as intercurrent illness, diet, and noncompliance with medication.

Forty subjects with a diagnosis of UCD who completed Study HPN-100-006 were enrolled.

Twenty additional UCD subjects ≥ 6 years of age were enrolled. These subjects included those who did not qualify for HPN-100-006 [e.g., subjects between the ages of 6-17; subjects with other UCD subtypes or adult subjects who have not taken sodium phenylbutyrate (NaPBA) in the past 6 months, etc.]. For adult subjects not receiving NaPBA in the past 6 months, subjects must, in the judgment of the investigator, be anticipated to benefit from the addition of a nitrogen-scavenging agent to their current treatment. See the inclusion criteria for examples of clinical evidence of potential benefit.

Monthly assessments included safety laboratory tests, amino acid panel, vital signs, electrocardiogram (ECG) monitoring, venous ammonia, and blood and urine metabolites. Adverse events (AEs) and concomitant medications were recorded on an ongoing basis.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who completed HPN-100-006:

  *Additionally, approximately 20 UCD subjects ≥ 6 years of age may be enrolled who have not participated in HPN-100-006. These subjects may include those who did not qualify HPN-100-006 (e.g., subjects between the ages of 6-17 years, subjects with other UCD subtypes, or adult subjects who have not taken sodium phenylbutyrate (NaPBA) in the past 6 months, etc.). For adult subjects not receiving NaPBA in the past 6 months, subjects must, in the judgment of the investigator, be anticipated to benefit from the addition of a nitrogen-scavenging agent to their current treatment. Clinical evidence of potential benefit from introduction of an ammonia-scavenging agent might include a recent history (in the past year) of clinically overt hyperammonemia accompanied by a venous ammonia ≥ 100 μmol/L, a recent history (within the past year) of protein intolerance, or a history of abnormally high venous ammonia levels accompanied by symptoms (e.g., headache) that might reasonably be attributed to hyperammonemia.
* Signed informed consent by subject and/or subject's legally acceptable representative.
* Diagnosis of urea cycle disorder (enzyme or transporter deficiency) confirmed via enzymatic, biochemical, or genetic testing.
* Able to perform and comply with study activities, including blood draws.
* Negative pregnancy test for all females of childbearing potential.
* All females of childbearing potential and all sexually active males must agree to use an acceptable method of contraception throughout the study.

Exclusion Criteria:

* Screening venous ammonia level of ≥ 100 μmol/L or signs and symptoms indicative of hyperammonemia; subjects may be re-screened after their venous ammonia is controlled, at the discretion of the investigator.
* History of 4 or more hyperammonemic events as defined in Section 3.5.1 in the preceding 12 months.
* Active infection (viral or bacterial) or any other condition that may increase venous ammonia levels.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
* Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication known to increase venous ammonia levels (e.g., valproate), within the 24 hours prior to Day 1 and throughout the study.
* History of QTc (QT interval corrected) prolongation, or a QTc interval ≥ 450 msec or an increase of ≥ 60 msec during the previous HPN-100 study if applicable.
* Known hypersensitivity to PAA or PBA.
* Liver transplant, including hepatocellular transplant.
* Breastfeeding or lactating females.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- United States (21):
  - Long Beach Memorial, Long Beach, California
  - UCLA, Los Angeles, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Univeristy of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - SNBL-Clinical Pharmacology Center, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944
- [Derived] Diaz GA, Krivitzky LS, Mokhtarani M, Rhead W, Bartley J, Feigenbaum A, Longo N, Berquist W, Berry SA, Gallagher R, Lichter-Konecki U, Bartholomew D, Harding CO, Cederbaum S, McCandless SE, Smith W, Vockley G, Bart SA, Korson MS, Kronn D, Zori R, Merritt JL 2nd, C S Nagamani S, Mauney J, Lemons C, Dickinson K, Moors TL, Coakley DF, Scharschmidt BF, Lee B. Ammonia control and neurocognitive outcome among urea cycle disorder patients treated with glycerol phenylbutyrate. Hepatology. 2013 Jun;57(6):2171-9. doi: 10.1002/hep.26058. Epub 2013 Jan 3. PMID 22961727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPN-100
Started | 60
Completed | 53
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | HPN-100
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.83 (13.933)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 54
  Canada | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adverse Events (Number of Participants Who Experienced Any AE Considered Related to Study Drug)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | HPN-100
Number analyzed (Participants) | 60
participants | 33

2. Secondary Outcome: Number and Causes of Hyperammonemic Events
Description: Number of hyperammonemic crises per patient
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: hyperammonemic events
Arm/Group | HPN-100
Number analyzed (Participants) | 60
hyperammonemic events | 0.20 (0.514)

3. Secondary Outcome: Blood Ammonia Levels
Description: Venous Ammonia levels over time
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: Umol/L
Arm/Group | HPN-100
Number analyzed (Participants) | 60
Umol/L
  Baseline | 27.623 (15.8875)
  Month 12 | 24.202 (20.6124)

4. Secondary Outcome: Patient Satisfaction With HPN-100
Description: Drug preference will be noted at week 3
Time Frame: Month 1 post dose
Population: all available questionnaires
Measure: Number; unit: % preferred HPN-100
Arm/Group | HPN-100
Number analyzed (Participants) | 50
% preferred HPN-100 | 90

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | HPN-100
Serious Adverse Events (participants affected / at risk) | 12/60
Other Adverse Events (participants affected / at risk) | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=60)
Abdominal pain (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 9
Dizziness (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=60)
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (General disorders) | 6
Constipation (General disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 7
Pyrexia (General disorders) | 4
Bronchitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis viral (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 19
Aspartate aminotransferase increased (Investigations) | 3
Vitamin D decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 8
Hyperammonaemia (Metabolism and nutrition disorders) | 9
Increased appetite (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Convulsion (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 3
Metrorrhagia (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days